CLINICAL TRIAL: NCT03644901
Title: Investigating the Role of ABO Blood Group in the Response to the Nonsurgical Periodontal Treatment.
Brief Title: Assessment of Response to the Conventional Periodontal Treatment Based on the Blood Group Phenotypes.
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Perio-03-2018
Record Dates: First submitted 2018-08-02; First posted 2018-08-23 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Root Planing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients whose blood type is A: Applying nonsurgical periodontal treatment (scaling and root planning).
  Interventions: Procedure: nonsurgical periodontal treatment
- Patients whose blood type is B: Applying nonsurgical periodontal treatment (scaling and root planning).
  Interventions: Procedure: nonsurgical periodontal treatment
- Patients whose blood type is AB: Applying nonsurgical periodontal treatment (scaling and root planning).
  Interventions: Procedure: nonsurgical periodontal treatment
- Patients whose blood type is O: Applying nonsurgical periodontal treatment (scaling and root planning).
  Interventions: Procedure: nonsurgical periodontal treatment

INTERVENTIONS:
Procedure: nonsurgical periodontal treatment — patients will undergo nonsurgical periodontal treatment to reduce the relative attachment level and improve the probing depth. An initial session will be conducted to remove supra gingival plaque and calculus. another appointment is set to perform full moth scalling and root planing.
  Other Names: Conventional periodontal treatment; scalling and root planing

SUMMARY:
The aim of this study is to find out if one blood group phenotype is more responsive than the others to the nonsurgical periodontal treatment.

DETAILED DESCRIPTION:
To the best of our knowledge, this is the first (research) randomized clinical trial that assesses how patient respond to the nonsurgical periodontal treatment based on their blood group phenotype.

ELIGIBILITY:
Inclusion Criteria:

* systematically healthy.
* have at least 20 teeth excluding the third molars.
* had not received any periodontal treatment or antibiotic therapy for dental or medical reason 6 month prior to the study.
* diagnosed with generalized chronic periodontitis (>30% of the sites have probing depth ≥4), and a minimum of six teeth with probing depth of 5-6 mm.

Exclusion Criteria:

* smokers and alcoholics.
* pregnancy.
* history of a systematic disease such as diabetes, leukemia, epilepsy.
* participants who are unable to perform routine oral hygiene.
* use of orthodontic appliances.
* participants who are unable to perform routine oral hygiene.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from chronic periodontitis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Change in relative attachment level. | measures will be taken at baseline and after two months from treatment.
  the relative attachment level measures the length form the base of the periodontal pocket to a stent

SECONDARY OUTCOMES:
Change in periodontal probing depth. | measures will be taken at baseline and after two months from treatment.
  the distance between the gingival margin to the base of the periodontal pocket.
Change in gingival index | index will be taken at baseline and after two months from treatment.
  it is used to designate the level of the gingival inflammation.
Change in plaque Index | index will be taken at baseline and after two months from treatment.
  it is used to designate the level of plaque accumulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ammar Kouky, DDS MSc, Principal Investigator — PhD Student in Periododontics, University of Damascus Dental School, Damascus; Mohammad Monzer Alsabbagh, DDS MSc PhD, Study Chair — Associate Professor of Periodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Periodontics, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pai GP, Dayakar MM, Shaila M, Dayakar A. Correlation between "ABO" blood group phenotypes and periodontal disease: Prevalence in south Kanara district, Karnataka state, India. J Indian Soc Periodontol. 2012 Oct;16(4):519-23. doi: 10.4103/0972-124X.106892. PMID 23493096
- [Background] Demir T, Tezel A, Orbak R, Eltas A, Kara C, Kavrut F. The Effect of ABO Blood Types on Periodontal Status. Eur J Dent. 2007 Jul;1(3):139-43. PMID 19212557
- [Background] Gautam A, Mittal N, Singh TB, Srivastava R, Verma PK. Correlation of ABO Blood Group Phenotype and Rhesus Factor with Periodontal Disease: An Observational Study. Contemp Clin Dent. 2017 Apr-Jun;8(2):253-258. doi: 10.4103/ccd.ccd_307_17. PMID 28839412
- [Background] Wang W, Liu L, Wang Z, Wei M, He Q, Ling T, Cao Z, Zhang Y, Wang Q, Shi M. Impact of ABO blood group on the prognosis of patients undergoing surgery for esophageal cancer. BMC Surg. 2015 Sep 29;15:106. doi: 10.1186/s12893-015-0094-1. PMID 26420728
- [Background] Yu Q, Wang L, Zhang S, Feng T, Li L, Chen B, Chen M. The role of ABO blood groups in Crohn's disease and in monitoring response to infliximab treatment. Blood Transfus. 2016 Sep;14(5):460-4. doi: 10.2450/2016.0199-15. Epub 2016 Feb 24. PMID 27136434